CLINICAL TRIAL: NCT06025916
Title: Postpartum Hemorrhage Reduction With Oral Tranexamic Acid (PROTECT): a Multicenter Randomized Controlled Trial
Brief Title: Postpartum Hemorrhage Reduction With Oral Tranexamic Acid: a Clinical Trial
Acronym: PROTECT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other); University of Cape Town (Other)
Responsible Party: Principal Investigator, Margit Endler, M.D. Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-00327
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: PPH
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (Active Comparator): Will receive 20ml of tranexamic acid 100mg/ml at a timepoint when the cervix is dilated 6 cn (for multipara) and 8 cm for primipara
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Will receive 20ml of placebo solution, equivalent in appearance and taste to tranexamic acid solution but with no active ingredient, at a timepoint when the cervix is dilated 6 cn (for multipara) and 8 cm for primipara
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — 20 ml of oral solution TA (100mg/ml)
  Other Names: Cyklokapron

SUMMARY:
This is a multicentre randomized placebo-controlled double-blinded phase IV study among 1000 women in Sweden and South Africa on the effect of oral tranexamic acid on PPH after vaginal delivery. The main purpose of the study is to evaluate the effect of orally administered tranexamic acid (TA) compared to placebo on rate of postpartum hemorrhage (PPH) after vaginal birth. Participants will be randomized to receive either 20 ml (2g) of the investigational medicinal product (TA100mg/ml) or 20ml of a placebo solution during labor. Our main endpoint, assessed at 24 hours after delivery is PPH defined as blood loss >=500ml and assessed both by weight and pre-postpartum hemoglobin (Hb) decrease >10 units difference in vaginal deliveries.

This RCT was preceded by a pilot intervention, included in the current protocol, aiming to assess uptake of oral forms of Tranexamic acid (TA) during active labour. The study took place at Södersjukhuset, Stockholm, Sweden between December 2022 and February 2023 among 51 women ≥ 36 gestational weeks with planned vaginal delivery who were randomized 1:1:1:1 to receive two grams of TA as oral solution, tablets, effervescent tablets, or 1g of intravenous (IV) TA, near full cervical dilatation. Blood samples were taken 30, 60, 120, 240, 360, and 480 minutes after TA administration. Plasma concentration of TA was measured using Liquid Chromatography-Tandem Mass Spectrometry. Mean values were compared between groups using ANOVA. Our main outcomes measures were time-to-therapeutic level, therapeutic interval, and maximum plasma concentration of TA.

DETAILED DESCRIPTION:
Background Severe PPH is the leading cause of maternal death worldwide especially in developing countries. Preventing PPH before onset is of key importance because once bleeding starts it is difficult to control.Tranexamic acid (TA) is a well-established medication for treatment and prevention of heavy bleeding. Oral forms of TA are available over the counter in many settings. The effect of oral treatment in vaginal deliveries has however been little studied and is a stated research priority by the WHO. Oral TA is low-cost, stable at room temperature and easy to administer which makes it especially applicable to both low resource delivery settings and home- births.To prevent PPH, a therapeutic serum concentration of TA should coincide with the period immediately after delivery of the child, when the risk of PPH is greatest, meaning that TA should optimally be administered during the latter part of active labor.

The premises of the RCT are the following:

1. The effect of oral prophylactic TA on rate of PPH is insufficiently known
2. If oral TA is effective in preventing PPH, routine administration could reduce maternal morbidity significantly at low expense.

Methods Study population and inclusion criteria The study will include 1000 women planned for vaginal delivery at three study sites in Sweden (n=500) and two study sites in South Africa (n=500) during the period September 2023 to December 2026. Enrolled women will be ≥18 years, ≥36 gestational weeks, and planned for vaginal delivery. Women with known bleeding disorders, known allergy to TA, ongoing treatment for venous thrombosis, or inability to make an informed consent will be ineligible.

Setting and duration: The study will take place between September 2023 and December 2026 at three study sites in Sweden as well as Mowbray Maternity Hospital and Khayelitsha District Hospital in South Africa.

Recruitment and randomization We will recruit women during a routine or planned antenatal visit after 35 gestational weeks, or after admission to the delivery ward during the latency phase of labor or the early stages of labor.

Randomization will occur after a woman has been admitted to the labor ward with spontaneous onset of labor. Participants will be randomized to receive either 20 ml of the investigational medicinal product (TA) or 20ml of a placebo solution. The randomization sequence will be computer-generated by KTA (Karolinska Clinical Trial Alliance) and flasks with the IMP/placebo will be marked according to this sequence. Randomization will be 1:1 in permuted blocks of 10 to allow for block-sized deliveries to study sites. The placebo will be developed and manufactured by Apotek Produktion och Laboratorier (APL), Sweden, who will also supply the TA. Placebo and IMP flasks, in their randomization sequence will be transported in a temperature-validated delivery to a central laboratory in Cape Town through World Courier who specialises in research related distributions.

Intervention Our intervention consists of the oral self-intake of either 20 ml (2g) of oral solution of TA, 20 ml of placebo equivalent in appearance, odor and taste to the IMP, when the cervix is fully dilated.

Primary endpoints Weight-estimated rate of PPH (≥500ml)

Secondary endpoints Pre-postpartum Hb difference (g/L) ≥10 units Weight-estimated rate of severe PPH (≥1000ml) Mean blood loss (ml) Mean pre-postpartum Hb decrease (units Rate of blood transfusion (%) Feasibility (adherence to protocol) Acceptability of the treatment among participants and providers Thromboembolism up to 6 weeks postpartum

Study procedures Participants will experience three study procedures that would not necessarily occur had they not taken part in the study but all of which form part of routine care.

1. A blood sample (hemoglobin, EVF, MCV, MCH, MCHC, LPC, TPC) taken at admission
2. The oral intake of 20 ml IMP/placebo at full cervical dilatation
3. Weighing of total blood loss (which is routine in many delivery settings)
4. A blood sample including (hemoglobin, EVF, MCV, MCH, MCHC, LPC, TPC) taken after 24 hours (or prior to discharge should discharge occur before 24 hours)

ELIGIBILITY:
Inclusion Criteria:

Enrolled women will be ≥18 years, ≥36 gestational weeks, and planned for vaginal delivery. Women with known bleeding disorders, known allergy to TA, ongoing treatment for venous thrombosis, or inability to make an informed consent will be ineligible.

Exclusion Criteria:

Opposite of above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
PPH | 24 hours
  Proportion of participants with weight-assessed blood loss after delivery >/= 500ml

SECONDARY OUTCOMES:
Severe PPH | 24 hours
  Proportion of participants with blood loss after delivery >/= 1000ml
Blood transfusion | 72 hours
  Proportion of participants receiving blood transfusion after vaginal birth
Mean blood loss | 24 hours
  Mean blood loss after vaginal delivery (ml) among participants
Mean pre-post partal hemoglobin | 24 hours
  Mean pre-post partal hemoglobin difference (units) among participants
Pre-post partal hemoglobin | 24 hours
  Pre-post partal hemoglobin >/= 10 units among participants
Thromboembolism | 6 weeks after delivery
  Proportion of participants with thromboembolic event postpartum
Feasibility of intervention | As specified in protocol
  Proportion of participants taking TXA/placebo according to protocol
Acceptability for participants | Delivery and 24 hours after delivery
  Rate of no to minor discomfort upon administration of intervention (acceptability) among participants
Acceptability for providers | Delivery and 24 hours after delivery
  Rate of no to minor disruption caused by administration of intervention (acceptability) experienced by providers

CONTACTS AND LOCATIONS:
Overall Officials: Margit Endler, MD PhD, Associate Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Södersjukhuset (South General Hospital), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Anonymized research data will be made available upon reasonable request

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: South Africa (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT06025916/Prot_SAP_001.pdf
  • Study Protocol: Swedish Pilot study preceding RCT and Swedish RCT protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT06025916/Prot_002.pdf